CLINICAL TRIAL: NCT05458817
Title: Digital-technology Based Interventions on Treatment of Migraine.
Acronym: Migrevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tartu University Hospital (Other)
Collaborators: University of Tartu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20148
Record Dates: First submitted 2022-01-21; First posted 2022-07-14 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Migraine; Primary Headache Disorders
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Primary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 1. Digital diary (Experimental): 75 participants in the group
  Interventions: Other: digital platform
- 2. Paper diary (Active Comparator): 75 participants in the group
  Interventions: Other: digital platform
- 3. Digital: diary and headache nurse (Experimental): 75 participants in the group
  Interventions: Other: digital platform
- 4. Paper diary and conventional headache nurse (Active Comparator): 75 participants in the group
  Interventions: Other: digital platform
- 5. Digital: diary, headache nurse and clinal psychologist (Experimental): 75 participants in the group
  Interventions: Other: digital platform
- 6. Paper diary, conventional headache nurse and conventional clinical psychologist (Active Comparator): 75 participants in the group
  Interventions: Other: digital platform
- 7. Digital: diary, headache nurse, clinal psychologist and physiotherapist (Experimental): 75 participants in the group
  Interventions: Other: digital platform
- 8. Paper diary, conventional: headache nurse, clinal psychologist and physiotherapist (Active Comparator): 75 participants in the group
  Interventions: Other: digital platform

INTERVENTIONS:
Other: digital platform — Patients in the digital group complete the tests in the patient's mobile application and/or in the Internet-based research environment of the Institute of Psychology of the University of Tartu kaemus.psych.ut.ee. Patients and specialists of the control group fill in the tests and the satisfaction questionnaire in the kaemus.psych.ut.ee environment.

SUMMARY:
The main aim of the research: To develop an interdisciplinary treatment platform based on digital technology and test the operation and effectiveness of digital interventions in comparison with conventional multidisciplinary treatment or treatment standards (incl. Paper diary, nurse counseling, physiotherapy, cognitive-behavioral therapy).

DETAILED DESCRIPTION:
Aims and purpose:

The main aim of the research: To develop an interdisciplinary treatment platform based on digital technology and test the operation and effectiveness of digital interventions in comparison with conventional multidisciplinary treatment or treatment standards (incl. Paper diary, nurse counseling, physiotherapy, cognitive-behavioral therapy).

Sub-aims:

To evaluate the effectiveness of interventions based on digital technology and their impact on the quality of life, comparing them with the interventions or treatment standards performed by ordinary specialists.

Assess the applicability and accessibility of digital technology-based interventions in the healthcare system against a treatment standard.

Determine the profile of patients (demographic and clinical indicators). Identify restrictions on the use of digital interventions. Evaluate patient compliance, non-specific treatment factors such as therapeutic relationship, and treatment credibility against the treatment standard.

Evaluate patient satisfaction with treatment methods and impact on treatment outcomes.

Assess the satisfaction of professionals with the implementation of a digital multidisciplinary treatment platform in patients.

Assess the use and generalization of digitally acquired skills in everyday practice.

Determine if and how much clinical contact is needed for digital-based interventions to be effective.

Evaluate cost-effectiveness against the standard of treatment. Assess the willingness to pay for the use of an effective headache treatment platform.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed migraine, frequent episodic, headache days a month 8-14 days;
2. patient age 18-64 years;
3. very good command of the Estonian language both orally and in writing.

Exclusion Criteria:

1. headaches lasting less than 8 days and more than 14 days per month;
2. all other primary and/or secondary diagnoses of headache;
3. under the age of 18 or over 64;
4. currently severe depression;
5. psychotic disorders;
6. pregnancy and lactation;
7. severe somatic disease;
8. severe organic mental disorders;
9. other chronic pain;
10. addictive disorders.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
headache frequency | 3 months
  headache diary: number of headache days per month
headache frequency | 6 months
  headache diary: number of headache days per month
headache frequency | 9 months
  headache diary: number of headache days per month

SECONDARY OUTCOMES:
medication use | 3 months
  headache diary: number of headache days per month
medication use | 6 months
  headache diary: number of headache days per month
medication use | 9 months
  headache diary: number of headache days per month
The effect of headaches on everyday life | 3 months
  Headache Impact Test (HIT-6)
The effect of headaches on everyday life | 6 months
  Headache Impact Test (HIT-6)
The effect of headaches on everyday life | 9 months
  Headache Impact Test (HIT-6)
Pain acceptance Pain acceptance Pain acceptance | 3 months
  Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R)
Pain acceptance Pain acceptance Pain acceptance | 6 months
  Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R)
Pain acceptance Pain acceptance Pain acceptance | 9 months
  Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R)
Pain-related anxiety | 3 months
  Pain Anxiety Symptoms Scale (PASS)
Pain-related anxiety | 6 months
  Pain Anxiety Symptoms Scale (PASS)
Pain-related anxiety | 9 months
  Pain Anxiety Symptoms Scale (PASS)
Health related quality of life | 3 months
  EUROHIS-QOL 8-item index (shortened version of the World Health Organization Quality of Life Instrument-Abbreviated Version)
Health related quality of life | 6 months
  EUROHIS-QOL 8-item index (shortened version of the World Health Organization Quality of Life Instrument-Abbreviated Version)
Health related quality of life | 9 months
  EUROHIS-QOL 8-item index (shortened version of the World Health Organization Quality of Life Instrument-Abbreviated Version)
Patient satisfaction with treatment 1 | 3 months
  Headache Attributed Lost Time (HALT)
Patient satisfaction with treatment 2 | 3 months
  Headache Under-Response to Treatment (HURT)
Patient satisfaction with treatment 3 | 6 months
  Headache Attributed Lost Time (HALT)
Patient satisfaction with treatment 4 | 6 months
  Headache Under-Response to Treatment (HURT)
Patient satisfaction with treatment 5 | 9 months
  Headache Attributed Lost Time (HALT)
Patient satisfaction with treatment 6 | 9 months
  Headache Under-Response to Treatment (HURT)
Cost-effectiveness 1 | 9 months
  databases of the Estonian Health Insurance Fund, the Social Insurance Board and the Institute for Health Development (insurance costs per patient - sick leaves compensation)
Cost-effectiveness 2 | 9 months
  databases of the Estonian Health Insurance Fund, the Social Insurance Board and the Institute for Health Development (insurance costs per patient - medications reimbursement)
Patient's willingness to pay for headache treatment | 9 months
  Willingness to pay bidding game

CONTACTS AND LOCATIONS:
Overall Officials: Mark Braschinsky, MD, PhD, Principal Investigator — Tartu University Hospital
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No